CLINICAL TRIAL: NCT03034837
Title: Economic Evaluation of ART Sealant in Preventing Pit and Fissure Caries in Permanent First Molars in an Asia Population
Brief Title: Effectiveness and Economic Evaluation of Glass Ionomer Material Using as Dental Sealant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Liu Baoying, Dr., Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201503121
Record Dates: First submitted 2017-01-23; First posted 2017-01-27 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Glass Ionomer Cement; Cost-effectiveness; Pit and Fissure Caries (Disorder)
MeSH Terms: conditions — Van der Woude syndrome

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Resin sealant (Active Comparator): Sealing pit and fissures of the included permanent first molars using "SDI conseal f" resin sealant material once at the baseline of the study.
  Interventions: Drug: resin sealant
- ART sealant (Experimental): Sealing pit and fissures of the included permanent first molars using "3M ESPE KetacTM Molar Easymix" glass ionomer cement material once at the baseline of the study.
  Interventions: Drug: ART sealant

INTERVENTIONS:
Drug: resin sealant — Sealing the occlusal surface of the included molars using the market product of SDI conseal f once.
  Other Names: SDI conseal f
  Arms: Resin sealant
Drug: ART sealant — Sealing the occlusal surface of the included molars using the market product of 3M ESPE KetacTM Molar Easymix" glass ionomer cement once.
  Other Names: GIC sealant; 3M ESPE KetacTM Molar Easymix" glass ionomer cement
  Arms: ART sealant

SUMMARY:
Eruption of the first permanent molar is the earliest in our oral cavity, leading to a high occurrence of dental caries in its pits and fissures. Early prevention of pit and fissure caries in this tooth is therefore of great importance for the preservation of a healthy dentition in one's life long time.

It has been shown that sealing the occlusal surface with pit and fissure sealant is a highly effective method to prevent pit and fissure caries. It has also been shown that the performance of sealing pits and fissures by glass ionomer materia l (the high viscosity, classification type 2 GIC material) using finger press method used in the atraumatic restoration method is as significant as that of using the traditional resin sealant material and technique.

The purpose of this study is to evaluate the long-term cost-effectiveness performance of the two sealing materials in the prevention of pits and fissures caries in young permanent molars of schoolchildren in a dental public health program to be held in primary schools. The findings will provide valuable information for decision making on the election of proper material and method for use in dental public program, especially for child population in the rural or social-economically deprived areas.

DETAILED DESCRIPTION:
Primary school children will be recruited and cluster randomized into three groups. Baseline dental check-up will be conducted to all the recruited children and dental status will be recorded. Placement of resin sealant or sealant using the glass ionomer material to the eligible permanent first molars or providing of oral health education will be interventions to the three groups respecively according to the group allocation. All the interventions will be provided only once in this study, and the children will be followed for at least 24 months at an six month interval to motor the dental caries of the included permanent first molars. Cost-effectiveness of placement of resin sealant and glass ionomer sealant will be evaluated and reported.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy grade 1-2 school children
* with written parental consent
* with at least 1 sound and fully erupted permanent first molar

Exclusion Criteria:

* Can not cooperate with the treatment
* Can not obtain the child's parental consent

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 329 (Actual)
Dates: Start 2016-01; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
cost-effectiveness of sealing | 24-month
  the incrental cost-effectiveness ratio of different sealing material used in this study in preventing pit and fissure caries in the permanent molars.

CONTACTS AND LOCATIONS:
Overall Officials: Baoying Liu, PhD, Principal Investigator — Zhengzhou University
Locations (2):
- China (2):
  - Jianxinjie Primary School, Zhengzhou, Henan
  - Ruhelu Primary School, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No